CLINICAL TRIAL: NCT01629277
Title: An Open-label, Single-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy and Safety of 24-hour Closed-loop Glucose Control in Comparison With Conventional Subcutaneous Insulin Pump Treatment Simulating Non-compliant Behaviours in Adolescents With Type 1 Diabetes
Brief Title: Closing the Loop in Adolescents During Non-compliance Behaviours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Principal Research Associate, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN03
Record Dates: First submitted 2011-04-04; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop insulin delivery; Non-compliant behaviours during adolescence
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Subcutaneous insulin delivery will be administered according the standard insulin pump settings
  Interventions: Device: standard insulin pump
- Closed-loop (Experimental): Subcutaneous insulin delivery will be adjusted according to the computer-based algorithm advice, based on subcutaneous glucose readings
  Interventions: Device: Closed-loop

INTERVENTIONS:
Device: Closed-loop — Subcutaneous insulin delivery will be adjusted according to the computer-based algorithm advice, based on subcutaneous glucose readings
  Arms: Closed-loop
Device: standard insulin pump — Subcutaneous insulin delivery will be administered according the standard insulin pump settings
  Arms: Control

SUMMARY:
The ultimate goal of the investigators ongoing research is the development of a closed-loop system for insulin delivery, which can help people with type 1 diabetes (T1D) attain a tight glucose control avoiding the risk of hypoglycaemia. The main components of the system are a continuous glucose monitor (CGM), an insulin pump and a computer-based 'model-predictive algorithm', which computes the amount of insulin to be given by the insulin pump according to the CGM values. In the studies performed thus far the efficacy and safety of closed-loop glucose control was evaluated both overnight and over a prolonged period of time including the day-time in children and adolescents with T1D. The results showed that closed-loop improved control of blood glucose and prevented nocturnal hypoglycaemia, as compared to the conventional insulin pump therapy.

The objective of the current study is to test the performance of closed-loop further, by evaluating the system during common non-compliant behaviours in the administration of meal insulin doses in adolescents with T1D. This will pave the way for a more comprehensive use of closed loop systems to control glucose levels in T1D under various "real-life mimicking" common circumstances. The present study adopts an open-label, randomised, 2 period cross-over design whereby closed-loop insulin therapy will be compared with the conventional insulin pump therapy in 12 adolescents with T1D.

Participants aged 12 to 18 years will be randomised for two 24 hour studies in a clinical research facility, during which glucose levels will be controlled by either the computer-based closed-loop algorithm (intervention arm) or by conventional insulin pump therapy (control arm). On both occasions, participants will under-estimate and omit the meal-related insulin dose for the evening-meal and lunch, respectively. The study will take place at the Wellcome Trust Clinical Research Facility (WTCRF), Cambridge with participants recruited from paediatric diabetes clinics in England.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-18 years
* Type 1 diabetes diagnosed for > 1 year
* Insulin pump treatment for at least 3 months
* HbA1c between 8 and 12%
* Subject willing to perform reduction/omission of meal insulin boluses during clinical studies

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Physical or psychological disease likely to interfere with the normal conduct of the study
* Current treatment with drugs known to interfere with glucose metabolism
* Known or suspected allergy against insulin
* Subjects with clinical significant nephropathy, neuropathy or proliferative retinopathy
* Total daily insulin dose >= 2 IU/kg/day
* Pregnancy, planned pregnancy, or breast feeding

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome measure | 24 hours
  The primary outcome measure is time spent with plasma glucose concentration in the target range (3.9-10.0mmol/L) between 19:00 on Day 1 and 18:00 on Day 2 (23 hours), as obtained with closed-loop insulin delivery as compared with conventional insulin pump therapy.

SECONDARY OUTCOMES:
Secondary efficacy outcome measure | 24 hours
  Secondary outcomes will include:
  * Time spent with plasma glucose concentration above the target range (>10mmol/L) between 19:00 on Day 1 and 18:00 on Day 2 (23 hours).
  * Time spent with plasma glucose concentration below the target range (<3.9mmol/L) between 19:00 on Day 1 and 18:00 on Day 2 (23 hours).
  * Total and basal insulin delivery between 19:00 on Day 1 and 18:00 on Day 2 (23 hours).
  * CGM glucose levels between 19:00 on Day 1 and 18:00 on Day 2 (23 hours).
  * Overnight plasma glucose levels between 24:00 on Day 1 and 08:00 on Day 2 (8 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Wellcome Trust Clinical Research Facility, Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357